CLINICAL TRIAL: NCT06464952
Title: Structure and Function of Microbiome Change in Subjects With Cirrhosis and PTSD After Potato Starch or Cellulose Supplementation (RESIST-PTSD)
Brief Title: Microbiome Modulation With Prebiotics in PTSD and Cirrhosis
Acronym: RESIST-PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BAJAJ0036
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cirrhosis; PTSD
Keywords: microbiome; prebiotic; gut-brain; liver disease
MeSH Terms: conditions — Fibrosis; Stress Disorders, Post-Traumatic; Liver Diseases

STUDY DESIGN:
Intervention Model Description: RCT in patients with cirrhosis and PTSD focused on feasibility and safety
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant potato starch (Experimental)
  Interventions: Dietary Supplement: Resistant potato starch
- Cellulose (Active Comparator)
  Interventions: Dietary Supplement: Powdered cellulose

INTERVENTIONS:
Dietary Supplement: Resistant potato starch — Prebiotic
  Arms: Resistant potato starch
Dietary Supplement: Powdered cellulose — Active comparator
  Arms: Cellulose

SUMMARY:
Despite medical advancements, PTSD remains a major issue in Veterans1. Current treatment strategies have relatively poor adherence. In patients with PTSD and cirrhosis, there is greater cognitive impairment as well as changes in gut microbiome structure and function2,3. In addition, when there is concomitant cirrhosis, medication-related treatment options become even narrower from a safety and tolerability perspective and cognitive issues pertaining to cirrhosis could impact participation3. Changes in gut microbiome in Veterans with cirrhosis and PTSD compared to those with cirrhosis without PTSD is characterized by a greater relative expression of pathobionts and reduction in stool microbiome diversity with reduction in bacteria that produce beneficial short chain fatty acids (SCFA)2. Modulation of the gut microbiome in patients with cirrhosis and PTSD may be an important therapeutic target. In prior studies with cirrhosis alone, microbial modulation using diet, antibiotics such as rifaximin, probiotics, and fecal microbiota transplant have improved gut microbial diversity and clinical outcomes in some cases4,5. In patients with cirrhosis without PTSD and in patients with PTSD without cirrhosis there is emerging evidence regarding prebiotics and other forms of gut microbial modulation.

Prebiotics are such an example6. Prebiotics are natural fibers derived from carbohydrates and can be beneficial to gut microbiota (good bacteria in the gut)6. Resistant starches (RS) are dietary fiber prebiotics found naturally in many foods including potatoes, plantains, and legumes6,7. In addition to being highly accessible, RS have been shown to be well tolerated with few adverse reactions. While no studies of RS exist in PTSD + cirrhosis patients, a meta-analysis of RS in IBD has shown RS to be an effective treatment in both animal and clinical studies where improvements in clinical remission and reduced mucosal damage were found7. However, there is insufficient data regarding patients with PTSD and cirrhosis regarding gut microbial structure and function modulation with dietary supplements such as resistant starches. These starches can improve SCFA production in elderly subjects, which could in turn affect the gut-brain axis favorably8.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Ability to provide informed written consent
3. Cirrhosis diagnosis
4. Willing to comply with all study procedures and be available for the duration of the study.
5. Ability to take oral medication.
6. Willing to provide study-related samples
7. Meeting the PCL-5 definition of PTSD and have a chart diagnosis of PTSD made by a mental health provider

Exclusion Criteria:

1. Known SARS-CoV-2 infection in the last 60 days using medical records
2. Subjects identified as, or appearing to, lack consent capacity
3. Alcohol abuse (greater than 14 drinks per week for men and 7 drinks per week for women)
4. Active illicit drug use (marijuana is allowed)
5. Use of investigational drugs, biologics, or devices within 30 days prior to randomization.
6. Individuals who are pregnant, lactating or planning on becoming pregnant during the study
7. Diagnosed inflammatory bowel disease, Crohn's disease, or Celiac disease
8. Unstable psychiatric illness (psychosis)
9. Previous gastrointestinal surgery (colorectal surgery, gastric bypass, intestinal resection)
10. Use of other prebiotics, probiotics (including yogurt containing live probiotics), postbiotics, or other fiber supplements in the last 30 days
11. Systemic antibiotics in the last 30 days
12. Fecal microbiota transplant in the last 30 days
13. Active dysphagia
14. Allergies to any of the ingredients in assigned products
15. Use of anti-diarrheal agents, stool softeners, or immunomodulatory medications in the last 30 days.
16. On treatment for hepatic encephalopathy.
17. Any other factor, condition, or medication not listed above the Investigators believe will affect the response in the gut or the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome Alpha Diversity between groups | 8 weeks
  Shannon diversity at end of interventions between both groups

SECONDARY OUTCOMES:
Gut microbiome Alpha Diversity within groups at study end | 8 weeks
  Shannon diversity at end of interventions within each group
Gut microbiome Alpha Diversity within groups at mid-study | 4 weeks
  Shannon diversity at mid-study within each group
Serum bile acids | 8 weeks
  Bile acid levels in serum at end of study between groups
Serum bile acids | 8 weeks
  Bile acid levels in serum at end of study within groups compared to baseline
Serum short-chain fatty acid (SCFA) levels | 8 weeks
  SCFA levels in serum at end of study between groups
Stool short-chain fatty acid (SCFA) levels | 8 weeks
  SCFA levels in stool at end of study between groups
Serum short-chain fatty acid (SCFA) levels | 8 weeks
  SCFA levels in serum at end of study within groups compared to baseline
Stool short-chain fatty acid (SCFA) levels | 8 weeks
  SCFA levels in stool at end of study within groups compared to baseline
MELD score change within group | 8 weeks
  MELD score within groups compared to baseline
MELD score change between groups | 8 weeks
  MELD score between groups
Adherence on assigned therapy | 8 weeks
  Proportion of assigned therapy taken during the entire study between groups (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States